CLINICAL TRIAL: NCT03012503
Title: The Effect of Biofreeze on Post Manipulation Soreness in Patients With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Robert Topp, Professor, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-2355
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Five minutes before cervical manipulation, controls received a placebo gel applied to their neck.
  Interventions: Drug: Placebos
- Treatment (Experimental): Five minutes before cervical manipulation the treatment group received a menthol containing gel (Biofreeze®) applied to their neck.
  Interventions: Drug: BioFreeze

INTERVENTIONS:
Drug: BioFreeze — The estimated surface area of the average adult's neck is 350cm and the standard dose of Biofreeze® to achieve a clinically significant effect has been sited to be 1ml/200cm2 of skin surface area. Using this data approximately 1.75 ml of the assigned gel was applied to each participant's neck (posterior, anterior, left lateral and right lateral) by the same member of the research team, 5 minutes prior to an independent practitioner performing cervical manipulation on the participant.
  Arms: Treatment
Drug: Placebos — control gel with a similar packaging, texture, and scent as Brand X but without the active ingredient of menthol
  Arms: Control

SUMMARY:
Background: Neck pain effects a significant number of individuals and is commonly treated with chiropractic cervical manipulation. The temporary increases in neck pain following cervical manipulation may contribute to a lack of compliance with prescribed therapy that following this therapy which in turn commonly contributes to protracted symptoms. Topical menthol has previously been shown to decrease pain shortly following application. The purpose of this study was to determine if patients with mechanical neck pain who received topical menthol gel applied to their neck prior to cervical manipulation would have less pain and increased neck range of motion following cervical manipulation than patients who did not receive menthol.

Methods: Patients, mean ages 35 years old, with non-radicular mechanical neck pain were randomly assigned to a control (n=31) or a treatment (n=29) group. Five minutes before cervical manipulation, controls received a placebo gel applied to their neck while the treatment group received a menthol containing gel (Biofreeze®) applied to their neck. Participants rated their neck pain on a 10-point scale prior to gel application (Pre) and at one minute (T1), 10 minutes (T2), 20 minutes (T3), and 30 minutes (T4) post cervical manipulation. Six measures of neck range of motion were assessed prior to topical applications of gel and at T1 and T4. ANCOVA repeated measures were performed to compare pain ratings and neck range of motion following manipulation while controlling for Pre measures.

DETAILED DESCRIPTION:
Background: Neck pain effects a significant number of individuals and is commonly treated with chiropractic cervical manipulation. The temporary increases in neck pain following cervical manipulation may contribute to a lack of compliance with prescribed therapy that following this therapy which in turn commonly contributes to protracted symptoms. Topical menthol has previously been shown to decrease pain shortly following application. The purpose of this study was to determine if patients with mechanical neck pain who received topical menthol gel applied to their neck prior to cervical manipulation would have less pain and increased neck range of motion following cervical manipulation than patients who did not receive menthol.

Methods: Patients, mean ages 35 years old, with non-radicular mechanical neck pain were randomly assigned to a control (n=31) or a treatment (n=29) group. Five minutes before cervical manipulation, controls received a placebo gel applied to their neck while the treatment group received a menthol containing gel (Biofreeze®) applied to their neck. Participants rated their neck pain on a 10-point scale prior to gel application (Pre) and at one minute (T1), 10 minutes (T2), 20 minutes (T3), and 30 minutes (T4) post cervical manipulation. Six measures of neck range of motion were assessed prior to topical applications of gel and at T1 and T4. ANCOVA repeated measures were performed to compare pain ratings and neck range of motion following manipulation while controlling for Pre measures.

ELIGIBILITY:
Inclusion Criteria:

* Individuals were included in the study if they were between the ages of 18-65 years old, presented to their with initial clinic visit with non-radicular mechanical neck pain greater than 3 on a 1-10 pain scale, and were prescribed by the clinical staff to receive a cervical manipulation

Exclusion Criteria:

1. Patients not receiving a cervical manipulation
2. Patients with radicular signs and/or symptoms
3. Patients who did not consent to be in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain over 5 time points | Prior to gel application (Pre) and at one minute (T1), 10 minutes (T2), 20 minutes (T3), and 30 minutes (T4) post cervical manipulation
  Participants rated their neck pain on a 10-point scale

SECONDARY OUTCOMES:
neck range of motion | Prior to gel application (Pre) and at one minute (T1), and 30 minutes (T4) post cervical manipulation
  Six measures of neck range of motion were assessed in the sagittal, frontal, and horizontal planes using the Acumar DataCapture hand-held dual inclinometer. This device has demonstrated a high degree of reliability (.87 - .92) without requiring calibration 21. These assessments included the neck motions of flexion, extension, right side bending, left side bending, left rotation and right rotation.

IPD SHARING:
Plan to Share IPD: No
Through publication and/or requests to the PI